CLINICAL TRIAL: NCT05945745
Title: Molecular Landscape Analysis and Clinical Implications for SCLC
Brief Title: Molecular Analysis and Treatment Options of SCLC
Status: Recruiting | Type: Observational
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xiaomin Niu, Principal Investigator, Shanghai Chest Hospital
Other Study IDs: THORACIC004
Record Dates: First submitted 2023-07-06; First posted 2023-07-14 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Small-cell Lung Cancer; Small Cell Lung Cancer, Combined Type; Small Cell Lung Carcinoma; Small Cell Lung Cancer Extensive Stage; Small Cell Lung Cancer Limited Stage
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Drug Therapy; Immunotherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Chemotherapy — different treatments based on the molecular analysis
  Other Names: immunotherapy; targeted therapy

SUMMARY:
Small cell lung cancer (SCLC) is an aggressive disease that is characterized by rapid growth and the early development of metastases. Patients typically respond to initial chemotherapy but quickly experience relapse, resulting in a poor long-term outcome. Therapeutic innovations that substantially improve survival have historically been limited, and reliable, predictive biomarkers are lacking.

Ongoing research has advanced the understanding of molecular categories and the immunologic microenvironment of SCLC, which in turn has helped improve disease classification and staging. Considering the role of molecular alterations has not yet fully to be defined in the treatment of SCLC, there is an urgent recognition that molecular alterations in the SCLC are important to predict response and survival for novel therapies and ongoing clinical trials. Advances in research have revealed critical information regarding biologic characteristics of the disease, which may lead to the identification of vulnerabilities and the development of new therapies. Further research focused on identifying biomarkers and evaluating innovative therapies will be paramount to improving treatment outcomes for patients with SCLC.

In summary, identification of (genetic) biomarkers in SCLC is increasingly essential to perform molecular diagnostics and individualized treatments. This project aims to create a registry of patients with SCCL to further the characterization of molecular alterations and develop (novel) treatments based on the detection.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of SCLC
* 18 years of age or older
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Histologically proven diagnosis of non-SCLC

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants with SCLC are with the standard treatment and/or are enrolled in the clinical trials.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 20 years
  Collect detailed clinical information on patients with SCLC via the electronic medical records
Disease control rate (DCR) | 20 years
  Collect detailed clinical information on patients with SCLC via the electronic medical records
Progression-free survival (PFS) | 20 years
  Collect detailed clinical information on patients with SCLC via the electronic medical records

SECONDARY OUTCOMES:
Overall survival (OS) | 20 years
  Collect detailed clinical information on patients with SCLC via the electronic medical records

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided